CLINICAL TRIAL: NCT05674825
Title: An Open-label, Navigational Investigation of Profile-related Evidence Determining Individualized Cancer Therapy for Patients With Aggressive Malignancies and Poor Prognoses
Brief Title: Investigation of Profile-related Evidence Determining Individualized Cancer Therapy for Patients With Aggressive Malignancies and Poor Prognoses
Acronym: MCW I-PREDICT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Hui-Zi Chen, MD, PhD, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00045600
Record Dates: First submitted 2022-12-23; First posted 2023-01-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: metastatic disease; unresectable disease; advanced malignancies; molecular profile
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1: Targeted agent (Experimental): Subjects will be grouped into one of three study groups (Groups 1, 2, or 3) based on their disease status and history of prior cancer therapy. Group 1 subjects will comprise treatment naïve subjects with localized disease and (i) are eligible for neoadjuvant treatment, (ii) have unresectable disease, or (iii) are medically unfit for surgical resection.
  Interventions: Drug: Targeted agent
- Group 1: Standard of care agent (Experimental): Subjects will be grouped into one of three study groups (Groups 1, 2, or 3) based on their disease status and history of prior cancer therapy. Group 1 subjects will comprise treatment naïve subjects with localized disease and (i) are eligible for neoadjuvant treatment, (ii) have unresectable disease, or (iii) are medically unfit for surgical resection.
  Interventions: Drug: Standard of care agent
- Group 2: Targeted agent (Experimental): Subjects will be grouped into one of three study groups (Groups 1, 2, or 3) based on their disease status and history of prior cancer therapy. Group 2 will comprise treatment naïve subjects with metastatic disease.
  Interventions: Drug: Targeted agent
- Group 2: Standard of care agent (Experimental): Subjects will be grouped into one of three study groups (Groups 1, 2, or 3) based on their disease status and history of prior cancer therapy. Group 2 will comprise treatment naïve subjects with metastatic disease.
  Interventions: Drug: Standard of care agent
- Group 3: Targeted agent (Experimental): Subjects will be grouped into one of three study groups (Groups 1, 2, or 3) based on their disease status and history of prior cancer therapy. Group 3 will comprise subjects with metastatic or unresectable disease who have received at least one prior systemic therapy, whether matched or unmatched.
  Interventions: Drug: Targeted agent
- Group 3: Standard of care agent (Experimental): Subjects will be grouped into one of three study groups (Groups 1, 2, or 3) based on their disease status and history of prior cancer therapy. Group 3 will comprise subjects with metastatic or unresectable disease who have received at least one prior systemic therapy, whether matched or unmatched.
  Interventions: Drug: Standard of care agent

INTERVENTIONS:
Drug: Targeted agent — The Molecular Tumor Board (MTB) will suggest molecularly targeted "matched" treatment.
  Arms: Group 1: Targeted agent; Group 2: Targeted agent; Group 3: Targeted agent
Drug: Standard of care agent — Subjects will receive treating physician's choice of traditional systemic therapy treatment for their malignancy, defined by National Comprehensive Cancer Network (NCCN) guidelines and/or tumor board recommendation(s).
  Arms: Group 1: Standard of care agent; Group 2: Standard of care agent; Group 3: Standard of care agent

SUMMARY:
This is a prospective, open-label navigational investigation designed to evaluate the feasibility of using molecular profile-based evidence to determine individualized cancer therapy for patients with aggressive malignancies. This is a non-randomized, histology-agnostic trial. Although there will be a case mix of histologies, the investigators now know that individual histologies are composed of a heterogeneous mix of molecular alterations. It is not clear whether one case mix is better or worse than another. Thus, the investigators are testing a strategy of molecular matching that may apply across different cancers.

DETAILED DESCRIPTION:
Eligible and consented patients, if not already performed, will have their tumor tissues/blood molecularly profiled. Patients will be stratified into Group 1 (treatment naïve, localized/unresectable/medically unfit for surgery), Group 2 (treatment naïve, metastatic), and Group 3 (prior treated). Based on multiomic profiling, matched therapy, if available, will be recommended by the Molecular Tumor Board. Patients who receive the recommended matched therapy are designated to Arm A. Otherwise, those that receive the unmatched therapy (i.e., treating physician's choice of therapy) or have no molecular alterations are designated to Arm B. The study feasibility will be measured by the ability to enroll patients, the acceptable turnaround time and the actionable information obtained from multiomic profiling, and the viability of identifying and delivering the matched therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patient with aggressive solid malignancy must meet at least one of the following:

   1. Malignancy with ≥30% two-year cancer-associated mortality as estimated by the treating oncologist and one of the study investigators and/or, where appropriate, according to accepted data sets in the field (e.g., NCDB). Diseases include but are not limited to: ampullary carcinoma, appendiceal cancer, colorectal cancer (CRC), extrahepatic cholangiocarcinoma (EHCC), esophageal adenocarcinoma, gallbladder cancer (GBCA) gastric adenocarcinoma, head and neck cancer, hepatocellular carcinoma (HCC), intrahepatic cholangiocarcinoma (IHCC), melanoma, non-KIT gastrointestinal stromal tumor (GIST), non-small cell lung cancer (NSCLC), ovarian cancer, pancreatic ductal adenocarcinoma (PDAC), sarcoma (high-grade), small bowel adenocarcinoma (including duodenal), triple-negative breast cancer (TNBC), urothelial cancer
   2. Refused standard therapies, OR
   3. Cancer of unknown primary or a rare tumor (i.e., fewer than 4 cases per 100,000 per year) with no approved therapies.
3. Patient with aggressive solid malignancy irrespective of two-year mortality who, in the opinion of the investigator, has no treatment option expected to yield significant clinical benefit.
4. Patient must have at least one of the following for a diagnosis/disease status:

   1. Unresectable disease, as determined by a disease-appropriate multidisciplinary tumor board.
   2. Medically unfit for surgical resection but with an expected survival of > three months.
   3. Localized disease and are eligible for neoadjuvant treatment.
   4. Metastatic disease.
   5. Disease where no conventional therapy leads to a survival benefit > six months in the respective cohort and line of therapy for which the patient is otherwise eligible.
5. Patient is either:

   1. Treatment naïve for their newly diagnosed malignancy (for enrollment to Groups 1 or 2), or
   2. Status post one or more systemic therapy regimens, whether matched or unmatched (for enrollment to Group 3). Note: There are no limitations on the number of prior local therapies.
6. Patient must have measurable disease for malignancy: defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, positron emission tomography (PET) -CT, MRI, or calipers by clinical exam.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
8. New York Heart Association (NYHA) Functional Classification I-II
9. Adequate organ and marrow function as defined below:

   1. Absolute neutrophil count ≥ 1.0 x 109/L
   2. Platelet count ≥ 75 x 109/L
   3. Total bilirubin ≤ 2.0 x institution's upper limit of normal (ULN)
   4. Patients without underlying liver disease

      • alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 3 x institutional ULN
   5. Serum creatinine ≤ 2.0 x institution's ULN or 24-hour creatinine clearance ≥ 30 ml/min
10. At the time of treatment, patient should be off other anti-tumor agents for at least five half-lives of the agent or two weeks from the last day of treatment, whichever is shorter to enroll in Group 3. Patient must not have been treated with anti-tumor agents to enroll in Group 1 or Group 2. Patient must be off prior antibody therapy for at least three half-lives before starting treatment.
11. Able to swallow and retain oral medication, if needed.
12. If actionable or appropriate molecular profiling has not already been performed, patient must have or provide evaluable tissue and/or blood for molecular profiling. This could be obtained during the standard of care tumor diagnosis or tumor staging evaluation. Tissue and/or blood is to be procured based on clinical discretion and discussion with the patient.
13. Pregnancy It is not known what effects matched therapy has on human pregnancy or development of the embryo or fetus. Therefore, female subjects participating in this study should avoid becoming pregnant, and male subjects should avoid impregnating a female partner. Non-sterilized female subjects of reproductive age and male subjects should use effective methods of contraception through defined periods during and after study treatment as specified below.

    Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
    * Not a female of childbearing potential (FCBP), defined as all female patients that were not in post-menopause for at least one year or are surgically sterile, OR
    * An FCBP must have a negative serum pregnancy test and agree to use at least one form of pregnancy prevention during the study for at least one month after treatment discontinuation unless otherwise noted by the agent(s) USPI or IB, which the FCBP must follow.

    Male participants: A male participant, even if surgically sterilized (i.e., status post-vasectomy), must use a form of barrier pregnancy prevention approved by the investigator or treating physician during the study and for at least one month after treatment discontinuation and refrain from donating sperm during this period unless otherwise noted by the agent(s) U.S. Prescribing Information (USPI) or investigator's brochure (IB), which the male participant must follow.
14. Ability to understand a written informed consent document, and the willingness to sign it.
15. Patients presented at Molecular Tumor Board (MTB) up to two weeks prior to signing consent are eligible to be treated on study based on the MTB recommendations and do not need to be represented at MTB prior to starting therapy on trial (unless six months elapsed between consent and start of study treatment).

Exclusion Criteria:

A potential study subject who meets any of the following exclusion criteria is ineligible to participate in the study.

1. Two oncologists disagree on prognosis or resectability.
2. Severe or uncontrolled medical disorder that would, in the investigator's opinion, confound study analyses of treatment response (i.e., uncontrolled diabetes, chronic renal disease, chronic pulmonary disease or active, uncontrolled infection, psychiatric illness/social situations that would limit compliance with study requirements).
3. Is pregnant or breastfeeding or any patient with childbearing potential not using adequate pregnancy prevention.
4. Whole brain radiation or stereotactic radiotherapy to CNS metastases within 14 days prior to start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Matched treatment | 8 months
  The number of subjects who receive matched treatment based on multiomic profiling analysis and MTB recommendations.

SECONDARY OUTCOMES:
Actionable alterations | 8 months
  The number of subjects who have a genetic test result that can be matched with appropriate treatment that can target their specific mutation.
MTB recommended treatment | 8 months
  The number of subjects who receive the MTB recommended treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Zi Chen, MD, PhD, Principal Investigator — Medical College of Wisconsin; Razelle Kurzrock, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No